CLINICAL TRIAL: NCT05897294
Title: Use of Voriconazole Inhalation Powder for the Treatment of Pulmonary Aspergillosis
Brief Title: Voriconazole Inhalation Powder for the Treatment of Pulmonary Aspergillosis
Status: No longer available | Type: Expanded Access
Sponsor: TFF Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TFF-VE-001
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Invasive Pulmonary Aspergillosis; Allergic Bronchopulmonary Aspergillosis; Chronic Pulmonary Aspergillosis; Aspergillus Tracheobronchitis; Anastomotic Infection; Pulmonary Fungal Infection
Keywords: voriconazole; Pulmonary Aspergillosis
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis; Aspergillosis, Allergic Bronchopulmonary; Lung Diseases, Fungal; Pulmonary Aspergillosis

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Voriconazole Inhalation Powder — dry powder inhalation of voriconazole
  Other Names: TFF VORI

SUMMARY:
Voriconazole Inhalation Powder is available on an expanded access basis to patients with pulmonary aspergillosis for up to 12 weeks. Duration of treatment may be extended on a case-by-case basis depending on drug availability and after discussion with the Sponsor.

DETAILED DESCRIPTION:
The purpose of this expanded access protocol is to provide, upon the treating clinician's request and Sponsor assessment, Voriconazole Inhalation Powder to patients with pulmonary aspergillosis, or patients with other voriconazole-sensitive pulmonary fungal infections, who have limited or no other treatment options or who have had unfavorable response to adequate standard of care antifungal therapy including to oral or intravenous voriconazole.

Reporting of serious adverse events (SAE) and Adverse Events of Special Interest (AESI) are required under this expanded access protocol. Patient treatment and outcomes information are also intended to be gathered under this protocol to the extent feasible (e.g., disease progression/improvement after treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or older at screening.
2. Diagnosed with pulmonary aspergillosis including Invasive Pulmonary Aspergillosis (IPA), Chronic Pulmonary Aspergillosis (CPA), Allergic Bronchopulmonary Aspergillosis (ABPA), Aspergillus tracheobronchitis and Aspergillus bronchial anastomotic infection. Pulmonary infections with voriconazole sensitive fungi other than Aspergillus such as but not limited to scedosporium and fusarium are also allowed.
3. Patient has limited or no treatment options due to documented or anticipated intolerance, toxicity, contraindications, or lack of clinical response to SOC antifungal therapy, as advocated by the relevant regional treatment guidelines.
4. The treating clinician considers that the potential advantage of using Voriconazole Inhalation Powder outweighs the potential risks. In patients with disseminated fungal infection in addition to pulmonary infection, Voriconazole Inhalation Powder must be used as add-on therapy to the current SOC.
5. The Sponsor agrees that the benefit:risk assessment is favorable for the use of Voriconazole Inhalation Powder in the patient.
6. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at Screening (Visit 1) and a negative urine pregnancy test (UPT) prior to first dose. Sexually active WOCBP and male patients must agree to use highly effective birth control or abstinence until 3 months after last dose.
7. Patient succeeds in meeting training criteria on the use of the dry powder inhaler (DPI) and is willing and able to perform adequate inhalation technique for treatment duration in the opinion of the treating clinician or designee.
8. Patient provides informed consent and agrees to follow the treatment regimen and safety and outcomes assessments.

Exclusion Criteria:

1. Infection with fungi not responsive to voriconazole.
2. Pregnant or breastfeeding.
3. History or presence of hypersensitivity or idiosyncratic reaction to voriconazole or excipients in Voriconazole Inhalation Powder.
4. Patients with severe liver disease as defined by Child-Pugh Class C.
5. Patients who are eligible and are able to participate in a clinical trial of Voriconazole Inhalation Powder.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult